CLINICAL TRIAL: NCT05845450
Title: Window-of-opportunity Umbrella Platform Trial of Short-course Pre-operative Targeted Treatments in Patients With Molecularly Selected and Resectable Primary Colorectal Cancer: the UNICORN Study
Brief Title: Pre-operative Targeted Treatments in Molecularly Selected Resectable Colorectal Cancer (UNICORN)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNICORN
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer; Resectable Colorectal Carcinoma
Keywords: targeted treatment; molecular alterations; platform trial
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trastuzumab deruxtecan; durvalumab; Panitumumab; balstilimab; sotorasib; Nivolumab

STUDY DESIGN:
Intervention Model Description: Phase II, multicentre, single-arm, open-label, multi-cohort trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- Cohort 1: HER2 positive (Experimental): Patients selected for the presence of pMMR/MSS status and HER2 overexpression/amplification defined as HER2 IHC 3+ or IHC 2+/ISH+ will receive the HER2 directed ADC trastuzumab deruxtecan 5.4 mg/kg IV on day 1.
  After receiving the short-course preoperative treatment, patients will undergo standard radical surgery. After surgery, patients will receive adjuvant chemotherapy as per national and international guidelines and according to the suggestion of a central multidisciplinary team. Then, standard follow up will be started as per local guidelines.
  Interventions: Drug: Trastuzumab deruxtecan
- Cohort 2: POLE/D1 mutated with ultra-mutated status (>100 Mut/Megabase) (Experimental): Patients selected for the presence of a proof-read domain pathogenic mutation of POLE/D1 associated with ultra-mutated status will receive a short-course preoperative immunotherapy treatment with the anti-PDL-1 monoclonal antibody durvalumab 1500 mg IV on day 1.
  After receiving the short-course preoperative treatment, patients will undergo standard radical surgery. After surgery, patients will receive adjuvant chemotherapy as per national and international guidelines and according to the suggestion of a central multidisciplinary team. Then, standard follow up will be started as per local guidelines.
  Interventions: Drug: Durvalumab
- Cohort 3: EGFR-dependent (Experimental): Patients selected for the presence of pMMR/MSS status, RAS and BRAF wild type status, PRESSING negative status and left-sided primary cancer will receive treatment with the anti-EGFR agent panitumumab 6 mg/kg IV on days 1 and 15.
  After receiving the short-course preoperative treatment, patients will undergo standard radical surgery. After surgery, patients will receive adjuvant chemotherapy as per national and international guidelines and according to the suggestion of a central multidisciplinary team. Then, standard follow up will be started as per local guidelines.
  Interventions: Drug: Panitumumab
- Cohort 4: pMMR/MSS status (Experimental): Patients selected for the presence of pMMR/MSS status and absence of HER2 overexpression/amplification, absence of POLE/D1 proof-read domain pathogenic mutation associated with ultra-mutated status will receive a short-course preoperative treatment with the anti-CTLA4 antibody botensilimab 1 mg/kg on day 1.
  After receiving the short-course preoperative treatment, patients will undergo standard radical surgery. After surgery, patients will receive adjuvant chemotherapy as per national and international guidelines and according to the suggestion of a central multidisciplinary team. Then, standard follow up will be started as per local guidelines.
  Interventions: Drug: Botensilimab
- Cohort 5: pMMR/MSS status (Experimental): Patients selected for the presence of pMMR/MSS status and absence of HER2 overexpression/amplification, absence of POLE/D1 proof-read domain pathogenic mutation associated with ultra-mutated status will receive a short-course preoperative treatment with the anti-CTLA4 antibody botensilimab 1 mg/kg on day 1 plus the anti-PD-1 balstilimab 3 mg/kg on days 1 and 15
  After receiving the short-course preoperative treatment, patients will undergo standard radical surgery. After surgery, patients will receive adjuvant chemotherapy as per national and international guidelines and according to the suggestion of a central multidisciplinary team. Then, standard follow up will be started as per local guidelines.
  Interventions: Drug: Botensilimab; Drug: Balstilimab
- Cohort 6: dMMR/MSI-H status (Experimental): Patients selected for the presence of dMMR/MSI-H status and absence of POLE/D1 proof-read domain pathogenic mutation associated with ultra-mutated status will receive a short-course preoperative treatment with the anti-CTLA4 antibody botensilimab 1 mg/kg on day 1.
  After receiving the short-course preoperative treatment, patients will undergo standard radical surgery. After surgery, patients will receive adjuvant chemotherapy as per national and international guidelines and according to the suggestion of a central multidisciplinary team. Then, standard follow up will be started as per local guidelines.
  Interventions: Drug: Botensilimab
- Cohort 7: dMMR/MSI-H status (Experimental): Patients selected for the presence of dMMR/MSI-H status and absence of POLE/D1 proof-read domain pathogenic mutation associated with ultra-mutated status will receive a short-course preoperative treatment with the anti-CTLA4 antibody botensilimab 1 mg/kg on day 1 plus the anti-PD-1 balstilimab 3 mg/Kg on days 1 and 15.
  After receiving the short-course preoperative treatment, patients will undergo standard radical surgery. After surgery, patients will receive adjuvant chemotherapy as per national and international guidelines and according to the suggestion of a central multidisciplinary team. Then, standard follow up will be started as per local guidelines.
  Interventions: Drug: Botensilimab; Drug: Balstilimab
- Cohort 8: KRAS G12C mutated (Experimental): Patients selected for the presence of pMMR/MSS status and KRAS G12C mutation will receive a short-course preoperative targeted treatment with the KRAS G12C inhibitor sotorasib 960 mg orally once daily from day 1 to 28 plus the EGFR inhibitor panitumumab 6 mg/kg IV on days 1 and 15.
  Interventions: Drug: Panitumumab; Drug: Sotorasib
- Cohort 9: pMMR/MSS status (Experimental): Patients selected for the presence of pMMR/MSS status, absence of HER2 overexpression/amplification, absence of POLE/D1 proof-read domain pathogenic mutation associated with ultra-mutated status and absence of KRAS G12C status will receive a short-course preoperative targeted treatment with the anti-EP4 agent vorbipiprant.
  Interventions: Drug: Vorbipiprant
- Cohort 10: pMMR/MSS status (Experimental): Patients selected for the presence of pMMR/MSS status, absence of HER2 overexpression/amplification, absence of POLE/D1 proof-read domain pathogenic mutation associated with ultra-mutated status and absence of KRAS G12C status will receive a short-course preoperative targeted treatment with the anti-EP4 agent vorbipiprant plus the anti PD-1 antibody nivolumab.
  Interventions: Drug: Vorbipiprant; Drug: Nivolumab

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — trastuzumab deruxtecan 5.4 mg/kg IV on day 1
  Arms: Cohort 1: HER2 positive
Drug: Durvalumab — durvalumab 1500 mg IV on day 1
  Arms: Cohort 2: POLE/D1 mutated with ultra-mutated status (>100 Mut/Megabase)
Drug: Panitumumab — panitumumab 6 mg/kg IV on days 1 and 15
  Arms: Cohort 3: EGFR-dependent; Cohort 8: KRAS G12C mutated
Drug: Botensilimab — botensilimab 1 mg/kg on day 1
  Arms: Cohort 4: pMMR/MSS status; Cohort 5: pMMR/MSS status; Cohort 6: dMMR/MSI-H status; Cohort 7: dMMR/MSI-H status
Drug: Balstilimab — balstilimab 3 mg/Kg on days 1 and 15
  Arms: Cohort 5: pMMR/MSS status; Cohort 7: dMMR/MSI-H status
Drug: Sotorasib — sotorasib 960 mg orally once daily from day 1 to 28
  Arms: Cohort 8: KRAS G12C mutated
Drug: Vorbipiprant — vorbipiprant 90 mg orally bid from day 1 to 28
  Arms: Cohort 10: pMMR/MSS status; Cohort 9: pMMR/MSS status
Drug: Nivolumab — 240 mg IV on days 1 and 15
  Arms: Cohort 10: pMMR/MSS status

SUMMARY:
This is a window-of-opportunity umbrella platform trial enrolling non-metastatic resectable colorectal patients selected for the presence of a specific targetable molecular alteration. The study aims to test the activity of specific targeted agents/combinations given as a short-course pre-operative strategy, matched with the specific alteration detected, followed by standard of care surgery.

DETAILED DESCRIPTION:
Patients with histologically confirmed non metastatic, radiologically staged as cT3-4 colorectal cancer eligible for radical surgery will be centrally molecularly prescreened by means of next-generation sequencing, HER2 IHC +/- HER2 silver-in situ hybridization and MMR proteins IHC with the aim to identify the presence of selected targetable molecular profiles/alterations. Whenever a pre-specified molecular profile/alteration is identified, the patient will be eligible for the matching Cohort and, after enrollment, will receive a specific short-course preoperative targeted treatment.

A total of 14 patients will be enrolled in each pre-specified molecularly-identified Cohort, according to the review of a Molecular Tumor Board established by the Sponsor, that will specifically evaluate the occurring and co-occurring molecular alterations.

Cohort 1 - patients with pMMR/MSS status and HER2 overexpression/amplification will receive the HER2 directed ADC trastuzumab deruxtecan 5.4 mg/kg IV on day 1.

Cohort 2 - patients with POLE/D1 mutation with ultra-mutated status (>100Mut/Megabase) will receive the anti-PDL-1 monoclonal antibody durvalumab 1500 mg IV on day 1.

Cohort 3 - COMPLETED - patients with EGFR-dependent tumor (pMMR/MSS status, RAS and BRAF wild type status, PRESSING negative status and left-sided primary cancer) will receive the anti-EGFR agent panitumumab 6 mg/kg IV on days 1 and 15.

Cohort 4 - COMPLETED - patients with pMMR/MSS status and absence of HER2 overexpression/amplification, absence of POLE/D1 proof-read domain pathogenic mutation associated with ultra-mutated status will receive the anti-CTLA4 antibody botensilimab 1 mg/kg on day 1.

Cohort 5 (opened sequentially, after completion of Cohort 4) -COMPLETED - patients with pMMR/MSS status and absence of HER2 overexpression/amplification, absence of POLE/D1 proof-read domain pathogenic mutation associated with ultra-mutated status will receive the anti-CTLA4 antibody botensilimab 1 mg/kg on day 1 plus the anti-PD-1 balstilimab 3 mg/Kg on days 1 and 15.

Cohort 6 - COMPLETED - patients with dMMR/MSI-H status and absence of POLE/D1 proof-read domain pathogenic mutation associated with ultra-mutated status will receive the anti-CTLA4 antibody botensilimab 1 mg/kg on day 1.

Cohort 7 (opened sequentially, after completion of Cohort 6) - COMPLETED - patients with dMMR/MSI-H status and absence of POLE/D1 proof-read domain pathogenic mutation associated with ultra-mutated status will receive the anti-CTLA4 antibody botensilimab 1 mg/kg on day 1 plus the anti-PD-1 balstilimab 3 mg/Kg on days 1 and 15.

Cohort 8 - patients with pMMR/MSS status and KRAS G12C mutation will receive the KRAS G12C inhibitor sotorasib 960 mg orally once daily from day 1 to 28 plus the anti-EGFR inhibitor panitumumab 6 mg/kg IV on days 1 and 15.

Cohort 9 - patients selected for the presence of pMMR/MSS status and absence of HER-2 overexpression/amplification, absence of POLE/D1 proof-read domain pathogenic mutation associated with ultra-mutated status, absence of KRAS G12C mutated status, will receive a short-course preoperative treatment with the anti-EP4 oral agent vorbipiprant 90 mg bid from day 1 to day 28.

Cohort 10 - Patients selected for the presence of pMMR/MSS status and absence of HER-2 overexpression/amplification, absence of POLE/D1 proof-read domain pathogenic mutation associated with ultra-mutated status, absence of KRAS G12C mutated status, will receive a short-course preoperative treatment with the anti-EP4 oral agent vorbipiprant 90 mg bid from day 1 to day 28 plus the anti PD-1 antibody nivolumab 240 mg on days 1 and 15.

After receiving the pre-specified study treatment, patients will be submitted to radical surgery at day 35 +/- 5 days. After surgery, patients will receive standard adjuvant chemotherapy as per national and international guidelines and according to the suggestion of a central multidisciplinary team. Then, standard follow up will be started as per local guidelines. Baseline assessments include radiological imaging (chest-abdomen-pelvis CT scan with contrast or abdomen MRI with contrast plus thorax CT without contrast if indicated, pelvis MRI mandatory for rectal cancer, and 18-FDG-PET scan if clinically indicated). Tumor re-assessments will be performed immediately prior to surgery at week 4-5. Safety assessments include monitoring of adverse events, clinical laboratory tests (chemistry, hematology, coagulation and urinalysis), vital signs, physical examinations and ECG as applicable.

Health-care related quality of life analysis will be done thanks to the administration of patient-reported outcomes questionnaires (EORTC QLQ-C30, EORTC QLQ-CR29, Euro QoL EQ-5D-5L) at baseline, during pre-operative treatment and at restaging.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria

* Provide a signed and dated informed consent document.
* Age ≥ 18 years at time of informed consent.
* ECOG PS of 0 and 1.
* Histologically confirmed colorectal cancer adenocarcinoma that is judged as initially resectable with elective surgery aimed at radical intent with R0 margins as per multidisciplinary team assessment.
* Radiological stage cT3-4, N0-2, M0 using computed tomography (CT) as in the pivotal FOxTROT study.
* Patients with rectal cancer candidate for R0 resection, not requiring pre-operative radiotherapy based on multidisciplinary team assessment, with the following characteristics on high-resolution thin slice (3 mm) contrast-enhanced magnetic resonance imaging (MRI):

  * ≤ T3a defined at the MRI (perivisceral fat infiltration <2 mm) and clinical N0
  * Upper-medium, defined as tumors with distal margin ≥ 5 cm from the anal verge.
  * Absence of mesorectal fascia invasion, as defined as a distance ≥ 1 mm between tumor and the mesorectal fascia.
* Able to provide enough archival FFPE tumor specimen that is already available from initial diagnostic procedures for the purpose of molecular pre-screening.
* Presence of one of the selected molecular profile/alteration after central pre-screening and necessary for the assignment to a matching treatment cohort.
* No prior systemic treatment for colorectal cancer or neoadjuvant radiation therapy for rectal cancer.
* Adequate bone marrow function (absolute neutrophil count ≥ 1.5 × 109/L; platelet count ≥ 100 × 109/L; hemoglobin ≥ 9.0 g/dL)
* Adequate renal function characterized by serum creatinine ≤ 1.5 × upper limit of normal (ULN) or calculated by Cockroft-Gault formula or directly measured creatinine clearance ≥ 50 mL/min at screening.
* Adequate hepatic function (serum total bilirubin ≤ 1.5 × ULN and < 2 mg/dL. Note: Patients who have a total bilirubin level 1.5 × ULN will be allowed if their indirect bilirubin level is ≤ 1.5 × ULN; Alanine aminotransferase and/or aspartate aminotransferase ≤ 2.5 × ULN).
* Women of childbearing potential must have a negative blood pregnancy test at the baseline visit. For this trial, women of childbearing potential are defined as all women after puberty, unless they are postmenopausal for at least 12 months, are surgically sterile, or are sexually inactive. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
* Subjects and their partners must be willing to avoid pregnancy during the trial and until a specific time interval after the last trial treatment: 7 months for female and 4 for male patients after last dose of trastuzumab-deruxtecan, 3 months for durvalumab, botensilimab and balstilimab and 2 months for panitumumab. Male subjects with female partners of childbearing potential and female subjects of childbearing potential must, therefore, be willing to use adequate contraception as approved by the Investigator (barrier contraceptive measure or oral contraception).
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.

Specific inclusion criteria for each Cohort

COHORT 1: pMMR/MSS status and HER2-positive status and LVEF ≥ 50% within 28 days before enrolment, international normalised ratio or Prothrombin time and either partial thromboplastin or activated partial thromboplastin time ≤ 1.5 × ULN

COHORT 2: Proofread domain mutations in POLE or POLD1 associated with ultra-mutated status, i.e. tumor mutational burden >100 Mut/Mb.

COHORT 3: pMMR/MSS status and wild-type status for RAS and BRAF, absence of molecular predictors of resistance (PRESSING panel negative), Left-sided and rectal primary tumor location, according to the specific inclusion criterion regarding rectal tumors.

COHORT 4: pMMR/MSS status and absence of HER2 overexpression/amplification, absence of POLE/D1 proof-read domain pathogenic mutation associated with ultra-mutated status and absence of KRAS G12C mutation.

COHORT 5: pMMR/MSS status and absence of of HER2 overexpression/amplification, absence of POLE/D1 proof-read domain pathogenic mutation associated with ultra-mutated status.

COHORT 6: dMMR/MSI-H status and absence of POLE/D1 proof-read domain pathogenic mutation associated with ultra-mutated status.

COHORT 7: dMMR/MSI-H status and absence of POLE/D1 proof-read domain pathogenic mutation associated with ultra-mutated status.

COHORT 8: pMMR/MSS status and KRAS G12C mutation, absence of HER2 overexpression/amplification and wild-type status for BRAF.

COHORT 9: pMMR/MSS status and absence of of HER2 overexpression/amplification, absence of POLE/D1 proof-read domain pathogenic mutation associated with ultra-mutated status, absence of KRAS G12C mutation.

COHORT 10: pMMR/MSS status and absence of of HER2 overexpression/amplification, absence of POLE/D1 proof-read domain pathogenic mutation associated with ultra-mutated status, absence of KRAS G12C mutation.

Exclusion Criteria:

General exclusion criteria

* Distant metastases at any site, as defined by negativity of chest/abdomen/pelvis contrast-enhanced computed tomography (CT).
* Risk criteria for obstructing disease at radiology or endoscopy as defined in the pivotal FOxTROT study.
* Need to receive neoadjuvant radiation or chemoradiation in patients with rectal cancer.
* Patients with known hypersensitivity to the study drug of the assigned cohort or to its excipients or to drugs belonging to the same drug class.
* Previous or concurrent malignancy within 2 years of study entry.
* Impaired cardiovascular function or clinically significant cardiovascular diseases, including any of the following: history of acute myocardial infarction, acute coronary syndromes (including unstable angina, coronary artery bypass graft, coronary angioplasty or stenting) ≤ 6 months prior to start of study treatment; symptomatic congestive heart failure (i.e., Grade 2 or higher), history or current evidence of clinically significant cardiac arrhythmia and/or conduction abnormality ≤ 6 months prior to start of study treatment, except atrial fibrillation and paroxysmal supraventricular tachycardia.
* Known history of HIV infection.
* Active infection including tuberculosis, hepatitis B, hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible only in case of negativity of HBV DNA. Patients positive for hepatitis C (HCV) antibody are eligible only if PCR is negative for HCV RNA.
* Other severe acute or chronic diseases that may increase the risk associated with study participation or study drug administration or that may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient an inappropriate candidate for the study.
* Any psychiatric condition that would prohibit the understanding or rendering of informed consent and that would limit compliance with trial requirements.
* Women in pregnancy or lactation condition. Women with child-bearing potential or sexually-active men not willing to use adequate contraception during whole study period.
* Use of any disallowed drugs.

Specific exclusion criteria for each Cohort:

COHORT 1:

* Previous treatment with a DXd-containing ADC or any anti-HER2 agent.
* Has LVEF< 50% within 28 days before enrolment.
* Has a history of (non-infectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at Screening. (eg, pulmonary emboli within 3 months of the enrolment, severe asthma, severe chronic obstructive pulmonary disease [COPD], restrictive lung disease, pleural effusion, etc.).
* Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (eg, pulmonary emboli within 3 months of the enrolment, severe asthma, severe chronic obstructive pulmonary disease [COPD], restrictive lung disease, pleural effusion, etc.).
* Any autoimmune, connective tissue, or inflammatory disorders where there is documented, or a suspicion of, pulmonary involvement at the time of Screening.
* Prior pneumonectomy.
* Has substance abuse or any other medical conditions that may interfere with the subject's participation in the clinical study or evaluation of the clinical study results.
* Patients with a medical history of myocardial infarction within 6 months before randomization/enrolment, symptomatic congestive heart failure (CHF) (New York Heart Association Class II to IV), subjects with troponin levels above ULN at screening (as defined by the manufacturer), and without any myocardial related symptoms, should have a cardiologic consultation before enrollment to rule out myocardial infarction.
* Corrected QT interval (QTcF) prolongation to > 470 msec (females) or >450 msec (males) based on average of the screening triplicate12-lead ECG.
* A pleural effusion, ascites or pericardial effusion that requires drainage, peritoneal shunt, or Cell-free and Concentrated Ascites Reinfusion Therapy (CART).

COHORT 2, 4, 5, 6, 7 and 10:

* History of autoimmune diseases or history of bone marrow or organ transplantation that requires immunosuppressive therapy.
* History of active primary immunodeficiency.
* Any condition requiring systemic treatment with corticosteroids at doses equal or superior to 10 mg daily of prednisone or equivalents, or other immunosuppressive drugs within 14 days from the inclusion in the study.
* Administration of live vaccines within 4 weeks from the inclusion in the study. Note: patients, if enrolled, should not receive live vaccine while receiving study drug(s) and up to 30 days after the last dose of study drug(s).
* Prior treatment with anti-CTLA4, anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents.

COHORT 3 and 8

* History of interstitial lung disease (e.g. pneumonitis or pulmonary fibrosis) or evidence of interstitial lung disease on baseline chest CT scan.
* Magnesium below the LNL.
* Prior treatment with an EGFR inhibitor.

COHORT 8:

* Patients who are unable to take a drug by mouth or previous clinical conditions or surgical resection that may affect the absorption of the study drug.
* Use of CYP3A4 or P-gp substrates with a narrow therapeutic window within 14 days or 5 half-lives of the drug or its major active metabolite, whichever is longer.
* Use of any herbal medications/supplements.
* Tumors with KRAS, NRAS, HRAS, BRAF or PTPN11 (SHP2) mutations, except KRAS G12C.
* Prior treatment with a KRAS G12C inhibitor.

COHORT 9 and 10:

* Prior treatment with EP4 receptor antagonists.
* Inability to swallow medications.
* Presence of portal hypertension and/or oesophageal varices.
* Known severe gastritis, duodenal or gastric ulcer, or any other condition that may lead to bleeding or perforation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
major pathological response rate | 5 weeks
  percentage of patients, relative to the total of enrolled subjects in the intention-to-treat population for each cohort, who will achieve a pathological complete response (pCR), defined as 0 or less residual viable tumor in both the primary tumor bed and lymphnodes, or major response (pMR), defined as 10% or less residual viable tumor, as per central pathological review in each Cohort.

SECONDARY OUTCOMES:
Treatment safety | 5 weeks
  incidence of AE (including SAEs) in each cohort during the short-course pre-operative treatment, assessed according to National Cancer Institute Common Toxicity Criteria version 5.0 (NCI-CTCAE v5.0).
Overall Toxicity Rate | 5 weeks
  percentage of patients, relative to the total of enrolled subjects of each cohort, experiencing any grade AE, according to NCI-CTCAE v5.0, during the short-course pre-operative treatment
G3/4 Toxicity Rate | 5 weeks
  percentage of patients, relative to the total of enrolled subjects in each cohort, experiencing any specific adverse event of grade 3/4, according to NCI-CTCAE v5.0, during the short-course pre-operative treatment.
Surgical mortality | 10 weeks
  the incidence of death occurring within 30 days after surgery in each cohort
Surgical morbidity | 10 weeks
  the incidence of a new onset temporary or permanent disability observed within 30 days after surgery in each cohort
Surgical complications | 18 weeks
  Surgical complications graded according to the Clavien-Dindo Classification of Surgical Complications and evaluated up to 90 days after surgery
Quality of life - PRO EORTC-QLQ-C30 | 5 weeks
  Quality of life will be assessed through Patient reported outcomes (PRO) instrument. EORTC QLQ-C30 For questions 1-28 of EORTC QLQ-C30 a 4-point scale is used. It scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit")and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome. For the questions 29 and 30 of EORTC QLQ-C30 a 7-points scale is used. It scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Half points are not allowed. The range is 6. First of all, raw score has to be calculated with mean values. Afterwards linear transformation is performed to be comparable. More points are considered to have a better outcome.
Quality of life - PRO EORTC-QLQ-CR29 | 5 weeks
  Quality of life will be assessed through Patient reported outcomes (PRO) instrument. EORTC QLQ-CR29.
  For questions 31-59 of EORTC QLQ-CR29 a 4-point scale is used. It scores from 1 to 4: 1 ("Not at all"), 2 ("A little"),3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome.
Quality of life - PRO EuroQol EQ-5D-5L | 5 weeks
  Quality of life will be assessed through Patient reported outcomes (PRO) instrument. EuroQol EQ-5D-5L. The EQ-5D-5L uses for first 5 questions qualitative multiple choice answers with NO SCALE. For the last questions, a score from 0 to 100 indicates from the worst to the best outcome.
changes in systemic immunity | 5 weeks
  defined by the longitudinal analysis of the peripheral blood subpopulations including myeloid cells (including myeloid-derived suppressor cells), CD8+ and CD4+ T lymphocytes (including T regulatory and Th17 cells), their proliferation and activation/exhaustion state collected at different time points performed by multiparametric cytometry
correlation of pCR/pMR with ctDNA mutational profiles | 5 weeks
  The correlation of pCR/pMR with ctDNA mutational profiles and its clearance after the specific short-course preoperative targeted treatment will be assessed by using ultra-deep whole-exome sequencing with Unique Molecular Identifiers to evaluate with high accuracy the presence of ctDNA in longitudinally collected liquid biopsies.
radiogenomic or radiomic signatures | 5 weeks
  To investigate the prognostic and/or predictive impact of radiogenomic or radiomic signatures in specific molecular subgroups, the baseline imaging will be analyzed to predict specific molecular profiles in all pre-screened patients, while the matched pre- and post-treatment imaging will be analyzed to predict tumor heterogeneity and pathological response in each cohort.
microbiota | 5 weeks
  The prognostic and/or predictive value of microbiota in specific molecular subgroups will be defined by investigating the composition of the gut microbiome in stool samples collected at pre-screening and at the end of short-course pre-operative treatment, its impact on outcomes of populations of molecular interest and its influence on the local and systemic immune responses to specific short-course preoperative treatments in each cohort.

OTHER OUTCOMES:
Disease-free survival | 36 months
  time from enrollment to the first documentation of disease recurrence or death due to any cause, whichever occurs first. DFS will be censored on the date of the last follow-up visit documenting absence of disease for patients who are alive, on study and disease free at the time of the analysis.
Overall survival | 36 months
  Overall survival will be defined as the time from enrollment to the date of death due to any cause. For patients still alive at the time of analysis, the OS time will be censored on the last date the patients were known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Pietrantonio, MD, Principal Investigator — Fondazione IRCCS - Istituto Nazionale dei Tumori di Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan, Lombardia/MI, Italy

IPD SHARING:
Plan to Share IPD: No
The trial results concerning the primary, secondary and exploratory outcomes will be published according to the standard guidelines. IPD could eventually be requested to the Sponsor and Principal Investigator, who will carefully evaluate the formal and motivated request